CLINICAL TRIAL: NCT06402097
Title: 'Transdermal Rigidity Assessment Via Ischemia of the Penis (TRIP). A New Sensor-driven Device to Measure Maximal Rigidity.'
Brief Title: TRIP-patch vs Duplex
Status: Completed | Type: Observational
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, Evelien Trip, Study Principal Investigator, St. Antonius Hospital
Other Study IDs: 70945
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Erectile Dysfunction
Keywords: rigiscan; erectile dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To measure saturation and desaturation of the cavernosal tissue with a cutaneous placed penile sensor, before and during full rigidity. To validate discriminating sensor-readings between flaccid state and full rigidity of the penis

DETAILED DESCRIPTION:
To measure saturation and desaturation of the cavernosal tissue with a cutaneous placed penile sensor, before and during full rigidity. To validate discriminating sensor-readings between flaccid state and full rigidity of the penis

ELIGIBILITY:
Inclusion Criteria:

* Indication for a penile duplex in our andrology clinic Signed informed consent Male Between 18-60 year

Exclusion Criteria:

* Patients who are unwilling to sign written informed consent
* Patients unable to undergo a duplex of the penis
* Patients with sickle cell anemia because this could affect the accuracy of the measurements

Ages: 18 Years to 60 Years | Sex: Male
Age Groups: Adult
Study Population: Patients with ED
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
change in sensor-readings | 1 hour
  To validate discriminating sensor-readings between flaccid state and full rigidity of the penis

CONTACTS AND LOCATIONS:
Locations (1):
- St Antonius Hospital, Nieuwegein, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No